CLINICAL TRIAL: NCT06513286
Title: TherVacB - A Multi-center Phase 1b/2a Trial to Assess Safety, Tolerability and Immunogenicity of a Heterologous Protein Prime/MVA Boost Therapeutic Hepatitis B Vaccine Candidate
Brief Title: TherVacB - A Heterologous Protein Prime/MVA Boost Therapeutic Hepatitis B Vaccine Candidate
Acronym: TherVacB
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: Institute of Virology Helmholtz Zentrum München Trogerstraße 30 81675 Munich, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Professor Dr. M. Hoelscher, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TherVacB_1b2a_1
Record Dates: First submitted 2024-06-11; First posted 2024-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm A1 (Experimental): HEPLISAV B® (low dose) and MVA-HBVac (low dose)
  Interventions: Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac)
- Arm A2 (Experimental): HEPLISAV B® (low dose) & HBcoreAg (low dose) and MVA-HBVac (low dose)
  Interventions: Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac)
- Arm A3 (Experimental): HEPLISAV B® (low dose) & HBcoreAg (low dose) and MVA-HBVac (high dose)
  Interventions: Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac)
- Arm A4 (Experimental): HEPLISAV B® (low dose) & HBcoreAg (medium dose) and MVA-HBVac (high dose)
  Interventions: Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac)
- Arm A5 (Europe) (Experimental): HEPLISAV B® (low dose) & HBcoreAg (low dose) and MVA-HBVac (high dose) or HEPLISAV B® (low dose) & HBcoreAg (medium dose) and MVA-HBVac (high dose)
  Interventions: Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac)
- Arm A6 (Tanzania) (Experimental): HEPLISAV B® (low dose) & HBcoreAg (low dose) and MVA-HBVac (high dose) or HEPLISAV B® (low dose) & HBcoreAg (medium dose) and MVA-HBVac (high dose)
  Interventions: Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac)
- Arm B1 (Experimental): HEPLISAV B® (high dose) & HBcoreAg (high dose) and MVA-HBVac (high dose)
  Interventions: Biological: TherVacB (2xHEPLISAV B + HBcoreAg + MVA-HBVac)
- Arm B2 (Experimental): HEPLISAV B® (high dose) & HBcoreAg (high dose) and MVA-HBVac (high dose) or regimen of study arm A5
  Interventions: Biological: TherVacB (2xHEPLISAV B + HBcoreAg + MVA-HBVac)

INTERVENTIONS:
Biological: TherVacB (HEPLISAV B +/- HBcoreAg + MVA-HBVac) — Administration of the described combinations via the intramuscular route
  Arms: Arm A1; Arm A2; Arm A3; Arm A4; Arm A5 (Europe); Arm A6 (Tanzania)
Biological: TherVacB (2xHEPLISAV B + HBcoreAg + MVA-HBVac) — Administration of the described combinations via the intramuscular route
  Arms: Arm B1; Arm B2

SUMMARY:
This study is an open-label, ascending dose phase 1b/2a trial to assess the safety and immunogenicity of a heterologous protein prime/MVA boost therapeutic hepatitis B vaccine in patients with chronic HBV who are virally suppressed with oral anti-viral therapies.

DETAILED DESCRIPTION:
This is a multi-centre study conducted in 81 participants. The clinical trial is divided into two overlapping parts (part A and B).

All treatment groups of Part A will receive a single dose of HEPLISAV B on Day 1 and Day 29 and MVA-HBVac on Day 56. From study arm A2 on all participants also receive HBcoreAg, in a low dose in arms A2 and A3 and in a medium dose in arm A4. In arms A5 and A6 either the low or the medium dose will be applied to an extended number of participants. The MVA-HBVac booster dose will be given in a dose-escalating way with a low dose in arms A1 and A2 and a high dose in arms A3, A4, A5 and A6.

The treatment group in Part B, study arm B1 will receive two doses of HEPLISAV B together with HBcoreAg in a high dose (on day 1 and 29), and a high booster dose of MVA-HBVac on day 56. In arm B2 either the regimen of B1 or A5 will be applied to an extended number of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the subject information and to personally name, sign and date the informed consent to participate in the clinical trial.
2. Provided written informed consent.
3. Confirmed chronic hepatitis B virus (HBV) infection (CHB) that fulfills the following criteria:

   * HBsAg positive for ≥ 6 months
   * Anti-HBs negative
   * HBsAg levels 100-2000 IU/mL
   * HBV nucleos(t)ide analog (NUC) treatment for ≥ 6 months
   * HBV load < 100 IU/ml at least twice within the last 6 months
4. Males and non-pregnant, non-lactating female with negative pregnancy test aged 18-70 years at time of informed consent.
5. Apart from CHB no other clinically significant health problems as determined during medical history and physical examination and clinical laboratory results at the screening visit. The following abnormal laboratory parameters will be permitted:

   * leukocyte count ≥ 2.500/µl
   * platelet count ≥ 150.000/µl
   * ALT elevation ≤ 60 U/L
   * AST should be ≤ 40 U/L
   * bilirubin should be ≤ ULN
   * INR should be ≤ ULN
   * CrCL > 60mL/min Non-clinically significant, minor deviations of laboratory measurements can be tolerated as they will not increase the risk of the individual having an adverse outcome from participating in this clinical trial as judged by the investigator.
6. Subject may be on chronic or as needed medications if, in the opinion of the investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate worsening of a pre-existing medical condition.
7. Body mass index 18.5-32.0 kg/m2 and weight >50 kg at screening.

Exclusion Criteria:

1. Known liver disease other than hepatitis B
2. Advanced liver fibrosis or cirrhosis (demonstrated by ultrasound or transient elastography ≥8 kP in fasting condition)
3. WOCBP who don't agree to comply with the applicable contraceptive requirements of the protocol
4. History of hepatocellular carcinoma
5. Coinfection with Hepatitis C Virus (HCV) (RNA positive), Human Immunodeficiency Virus (HIV) or Hepatitis Delta virus (anti-Delta positive)
6. Regular alcohol intake >30 g/d (male), >20 g/d (female) or any other known drug addiction.
7. Donation of blood or blood products (e.g., 450 mL or more of plasma or platelets) within 60 days prior to receiving the first dose of the investigational medicinal product (IMP).
8. Receipt of any vaccine in the 2 weeks prior to first trial vaccination (4 weeks for live vaccines), during trial or planned receipt of any vaccine in the 3 weeks following last trial vaccination. Exception: Required recommended pandemic vaccines or emergency vaccines (e.g., tetanus) are allowed.
9. Previous receipt of an MVA based vaccine (e.g. as part of previous MVA studies, monkeypox or smallpox vaccination)
10. Known allergy to components of the vaccine products as referred in Table 6 (incl. hypersensitivity to yeast components, E.coli proteins or lipids, duck's or hen's egg white, penicillin, streptomycin, , kanamycin) or history of life-threatening reactions to vaccines containing one of the substances.
11. Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccines.
12. Clinically relevant findings in ECG or significant thromboembolic events in medical history.
13. Evidence for a condition in the subject's medical history or during medical examination that might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of vaccine products.
14. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the first dose of the trial vaccine.
15. Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 3 years.
16. Any treatment with immunosuppressants or other immune-modifying drugs (including, but not limited to systemic corticosteroids, biologicals and Methotrexate) within the last 3 years. Exception: topical corticosteroids, e.g. occasional asthma spays or systemic corticosteroids for medical emergencies.
17. Any chronic or active neurologic disorder, including diagnosis of migraine, seizures and epilepsy. Exception: a febrile seizure as a child and occasional headaches.
18. Participation in a clinical investigation within the past 4 weeks or five times the half-life of the previously taken IMP.
19. Investigator or employee of the study site with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, natural or adopted child) of the investigator or employee with direct involvement in the proposed study.
20. Subjects who are known or suspected

    * not to comply with the clinical trial directives.
    * not to be reliable or trustworthy.
    * not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequencies and magnitudes of unsolicited adverse events | up to day 84
  Reported numbers and severity grade of unsolicited AEs for 28 days after each vaccination
Frequencies and magnitudes of serious adverse events (SAEs) throughout the trial period | up to day 224
  Reported numbers and types of SAEs throughout the period of the clinical trial
Frequencies and magnitudes of adverse event of special interest (AESI) and Suspected Unexpected Serious Adverse Reaction (SUSAR) throughout the trial period | up to day 224
  Reported numbers and severity grade of AESIs and numbers and types of SUSARs
Frequencies and magnitudes of solicited local reactogenicity signs and symptoms within 7 days after each vaccination | up to day 63
  Reported numbers and severity of solicited AEs
Frequencies and magnitudes of solicited systemic reactogenicity signs and symptoms within 7 days after each vaccination | up to day 63
  Reported numbers and severity of solicited AEs
Frequencies and magnitudes of liver toxicity (ALT flare-ups) stratified by severity throughout the trial period | up to day 224
  Reported numbers and severity grade of AESIs
Change from baseline of safety laboratory measurements throughout the trial period | up to day 224
  Changes of values from safety laboratory measurements from baseline

SECONDARY OUTCOMES:
Frequency of subjects with HBsAg drop below the lower limit of quantification | 2 weeks (Day 70), 2 months (Day 112) and 6 months (Day 224) after completion of the vaccination regimen (last study visit).
  Determined by an accredited serological immuno-assay
Frequency of subjects with a ≥ 1 log10 drop in HBsAg titers from day 0 (start of study medication) with the goal of 30% of patients achieving a ≥ 1log10 HBsAg drop | 2 weeks (Day 70), 2 months (Day 112) and 6 months (Day 224) after completion of the vaccination regimen (last study visit
  Determined by an accredited serological immuno-assay
Frequency of subjects with an induction of anti-HBs titers ≥ 10 IU/L | 2 weeks (Day 70), 2 months (Day 112) and 6 months (Day 224) after completion of the vaccination regimen (last study visit
  Determined by an accredited serological immuno-assay
Frequency of subjects developing any anti-HBs antibody response | 2 weeks (Day 70), 2 months (Day 112) and 6 months (Day 224) after completion of the vaccination regimen (last study visit
  Determined by an accredited serological immuno-assay
Frequency of subjects with an increased signal in the HBV-specific cytokine-secretion assay compared to pretreatment values | 2 weeks (Day 70), 2 months (Day 112) and 6 months (Day 224) after completion of the vaccination regimen (last study visit
  Determined by cytokine release assays

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof. Dr. med., Study Chair — Division of Infectious Diseases and Tropical Medicine, LMU Klinikum
Locations (6):
- Germany (6):
  - Investigational Site GUF, Frankfurt
  - Investigational Site UKE, Hamburg
  - Investigational Site MHH, Hanover
  - Investigational Site Uni Leipzig, Leipzig
  - Investigational Site LMU, Munich
  - Investigational Site TUM, Munich

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan is in preparation